CLINICAL TRIAL: NCT01401309
Title: Effects of Respiratory Gating on FDG/PET Detection of Hepatic Metastasis in Patients With Colon Cancer
Brief Title: PET Respiratory Gating to Detect Hepatic Metastasis in Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: Southwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SRMC 10-07
Record Dates: First submitted 2011-01-24; First posted 2011-07-25 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to examine if there is improved sensitivity in detecting hepatic lesions using respiratory gating and if there is an improvement in confidence defining lesions as benign or malignant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colon cancer
* 18 years or older
* Signed Informed Consent Form
* Blood Glucose of 200 or less prior to scan

Exclusion Criteria:

* Patients with known hepatic metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Detecting | Jan 2011 - Nov 2011
  To exam if there is an improved sensitivity in detecting hepatic lesions using respiratory gating and if there is improvement in confidence defining lesions as benign or malignant

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Treamtent Centers of America at Southwestern Regional Medical Center, Inc, Tulsa, Oklahoma, United States